CLINICAL TRIAL: NCT03622164
Title: Randomized Trial of Unilateral vs. Bilateral Neck Irradiation in Head and Neck Cancer Patients Treated With Primary Surgery
Brief Title: Unilateral Neck Radiotherapy in Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0002
Record Dates: First submitted 2018-07-09; First posted 2018-08-09 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Neoplasms
Keywords: radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-experimental intervention (Active Comparator): Radiotherapy to the bilateral neck lymphatics and tumor bed (radiotherapy to both sides of the neck).
  Interventions: Radiation: Radiotherapy to the bilateral neck lymphatics and tumor bed (radiotherapy to both sides of the neck)
- Experimental intervention (Experimental): Radiotherapy to ipsilateral neck lymphatics and tumor bed (radiotherapy to one side of the neck).
  Interventions: Radiation: Radiotherapy to ipsilateral neck lymphatics and tumor bed (radiotherapy to one side of the neck)

INTERVENTIONS:
Radiation: Radiotherapy to ipsilateral neck lymphatics and tumor bed (radiotherapy to one side of the neck) — CTV54 includes only the ipsilateral neck, including levels 2-4 plus levels 1 and/or 5 as clinically indicated.
  Arms: Experimental intervention
Radiation: Radiotherapy to the bilateral neck lymphatics and tumor bed (radiotherapy to both sides of the neck) — CTV54 includes the entire surgical bed, including bilateral neck lymphatics at risk of harboring microscopic disease
  Arms: Non-experimental intervention

SUMMARY:
Patients with head and neck cancer typically undergo a surgical procedure to remove the lymph nodes that could contain disease on both sides of the neck. After surgery, radiotherapy is given (with or without chemotherapy) to the area that underwent surgery and both sides of the neck, even if disease was only found on one side. Giving radiotherapy to both sides of the neck commonly results in high rates of side effects, which in turn affects patient quality of life.

There is growing evidence from some other studies that support the safety of omitting radiotherapy after surgery in the side of the neck with no disease. With this study, the investigators are hoping to justify its routine use and, if successful, the standard of care could be to receive radiation on only one side of the neck instead of both sides. This could alleviate the extent of some side effects and improve patient quality of life.

Participants will be randomized into one of the following groups to receive radiotherapy as follows:

Arm 1 (Non-experimental intervention): standard intervention: Radiotherapy to both sides of the neck. Treatment will begin a maximum of 8 weeks from the surgery date.

Arm 2 (Experimental intervention): Radiotherapy to one side of the neck. Treatment will begin a maximum of 8 weeks from the surgery date.

ELIGIBILITY:
Inclusion Criteria:

Patients with squamous cell carcinoma of the head and neck undergoing primary surgical management are eligible to participate if they meet the following eligibility criteria:

* Age ≥18
* Primary site of disease in the oral cavity, oropharynx, larynx, or hypopharynx.
* Squamous cell carcinoma confirmed by histology.
* Bilateral modified radical or selective neck dissections carried out as part of primary surgery, with >= 10 lymph nodes removed from the contralateral neck
* The contralateral neck is pathologically negative
* Pre-surgical FDG-PET/CT scan did not show any clinically involved contralateral neck nodes.
* Patients must have the ability to read, understand, and sign an informed consent and must be willing to comply with study treatment and follow-up.

Exclusion Criteria:

* Previous radiation to the head and neck area
* Pregnancy
* Other contraindications to radiation treatment (e.g. severe connective tissue disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Locoregional control | At 24 months
  Locoregional failure is defined as disease recurrence (by imaging, clinical exam, or biopsy) in the neck or at the primary site.

SECONDARY OUTCOMES:
Overall survival and disease-specific survival | 5 years after diagnosis or the start of treatment.
  Percentage of people in a study or treatment group who are alive five years after their diagnosis or the start of treatment.
University of Washington Quality of Life Questionnaire - Radiation Therapy Oncology Group (UW-QOL - RTOG) modification | At 6, 12, 18 and 24 months post radiotherapy
  The University of Washington Quality of Life questionnaire Radiation Therapy Oncology Group (RTOG) modification, is a health related quality of life tool for use in head and neck cancer patients receiving RT.
  The UW-QOL RTOG modification consists of 15 items with response options ranging from 10 to 50, in multiples of 10. That is, the lowest symptom burden is rated as 10, whereas the highest symptom burden is rated as 50. The individual item scores are totaled and then averaged to obtain the final score. This scoring results in a lower score indicating greater HR-QOL; and conversely, higher scores indicating lower HRQOL.
Xerostomia | At 6, 12, 18 and 24 months post radiotherapy
  Overall score
Acute toxicity | Weekly throughout RT treatment (approximately 6 weeks)
  Toxicity scoring will be carried out to include salivary gland, mucositis, skin, and fatigue grading according the CTCAE version 4.0 scoring criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada